CLINICAL TRIAL: NCT03186014
Title: A Novel Fully Covered Segmented Irradiation Stent Loaded With 125I Seeds for the Palliation of Malignant Dysphagia：a Prospective Pilot Study
Brief Title: A Fully Covered Irradiation Stent for the Palliation of Malignant Dysphagia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Director of Department of Interventional Radiology & Vascular Surgery, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017ZDSYLL027
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Malignant Dysphagia
Keywords: Malignant dysphagia; Stent; Esophageal neoplasms; Brachytherapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fully covered irradiation stent (Experimental): A esophageal fully covered segmented irradiation stent loaded with 125I seeds is placed in Patients with malignant dysphagia
  Interventions: Device: Fully covered irradiation stent

INTERVENTIONS:
Device: Fully covered irradiation stent — A esophageal fully covered segmented irradiation stent loaded with 125I seeds is placed in Patients with malignant dysphagia

SUMMARY:
Dysphagia is the major symptom of patients with malignant esophageal stricture caused predominantly by advanced esophageal cancer. Stent placement is the most commonly used strategies for relieving the dysphagia and a novel irradiation stent loaded with 125I seeds has recently been developed. A multicentre randomized clinical trial demonstrated this irradiation stent can relieve the dysphagia rapidly and prolong the survival of patients with advanced esophageal cancer, but the total stent stenosis rate cannot be ruduced. A novel fully covered segmented retrievable irradiation stent was developed in our institute. The purpose of this study is to evaluate the safety and clinical efficacy of this newly developed irradiation stent in patients with unresectable malignant dysphagia.

DETAILED DESCRIPTION:
Esophageal cancer is the eighth most common cancer and the sixth leading cause of cancer related mortality worldwide. Most patients have lost chance of surgical resection when they are initially diagnosed, because of late stage cancer or metastasis. Dysphagia is the major symptom of patients with advanced esophageal cancer. The two most commonly used strategies for relieving the dysphagia are stent placement and intraluminal brachytherapy. Stent placement provides a fast improvement of dysphagia, while intraluminal brachytherapy provides a more durable effect on dysphagia. To combine the advantages of the immediate relief of esophageal dysphagia with stent placement and long-term benefit with brachytherapy, a novel irradiation stent loaded with 125I seeds has been developed in the authors' institute. Recently, a multicentre randomized clinical trial demonstrated this novel irradiation stent can relieve the dysphagia rapidly and prolong the survival of patients with advanced esophageal cancer. However, this irradiation stent only provides a slightly longer relief of dysphagia and cannot reduce the total stent stenosis rate, because partly covered stent with uncoated flanges on both ends for anchoring the stent are used. In the past few years, fully covered retrievable stents which allow less tissue overgrowth have been used in patients with longer life expectancy, especially if they are receiving additional palliative therapy like brachytherapy. In order to provide a further longer relief of dysphagia and prevent stent migration caused by tumor regresses with brachytherapy, a fully covered segmented retrievable irradiation stent has been developed. The aim of the current study is to evaluate the clinical efficacy, particularly focus on stent stenosis and stent migration, and safety of this newly developed irradiation stent in patients with unresectable malignant dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopically and histologically confirmed malignant obstruction of the esophagus or the gastroesophageal junction
* Progressive dysphagia with a dysphagia score of 2-4
* Unresectable tumours due to extensive lesions, metastases, or poor medical condition
* Patients with clear consciousness, cooperation
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-3
* Informed consent: authorization and signature

Exclusion Criteria:

* The superior border of the lesion extending beyond the level of the seventh cervical vertebrae
* Previous treatment with a stent or surgical resection for the same condition
* Ulcerative esophageal cancer
* Esophageal fistula
* Severe hepatic inadequacy or renal inadequacy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Recurrent dysphagia | Participants will be followed till die or lost to follow-up, an expected average of 6 months.
  The rate of occurrence of tissue ingrowth or overgrowth, stent migration, and food obstruction.

SECONDARY OUTCOMES:
Dysphagia score | Baseline, post-op 7 days, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months
  Investigated with the Ogilvie score: 0 for nil, 1 for normal diet avoiding certain foods such as raw apple and steak, 2 for semi-solid diet, 3 for fluids only, and 4 for complete dysphagia, even for liquids.
ECOG performance status | Baseline, post-op 7 days, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months
  Utilizing ECOG performance status score to assess the functional status.
EORTC QLQ-C30 | Baseline, post-op 7 days, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months
  Utilizing EORTC QLQ-C30 to assess the health-related quility of life.
EORTC QLQ-OG25 | Baseline, post-op 7 days, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months
  Utilizing EORTC QLQ-OG25 to assess the health-related quility of life in patients with cancer of the oesophagus and the oesophago-gastric junction.
Technical success | During operation
  The rate of adequate placement of the stent in the target position and good passage of contrast medium through the stent into the stomach.
Clinical success | 3 days after stent placement
  The rate of relief of dysphagia with a decrease of at least one point in the dysphagia score.
Overall survival | Participants will be followed till die or lost to follow-up, an expected average of 6 months.
  Time from initial stenting to the day when the patients died or lost to follow-up.
Stent patency | Participants will be followed till die or lost to follow-up, an expected average of 6 months.
  Time from initial stenting to the day when recurrent dysphagia occured or patients died.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Participants will be followed till die or lost to follow-up, an expected average of 6 months.
  Adverse events including hemorrhage, perforation, fistula, severe chest pain, and pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-jun Teng, Ph.D,MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital,Southeast University, Nanjing, Jiangsu, China